CLINICAL TRIAL: NCT01257620
Title: Exploratory, Randomized, Double-blind, Placebo-Controlled Study on the Effects of Bifidobacterium Infantis in Active Celiac Disease
Brief Title: Clinical Trial on the Effects of Bifidobacterium Infantis in Active Celiac Disease
Acronym: Celiac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bai, Julio M.D. (Individual)
Collaborators: The National Institute of Probiotics (Other)
Responsible Party: Principal Investigator, Bai, Julio M.D., Principle Investigator, Dr. C. Bonorino Udaondo Gastroenterology Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Celiac
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Celiac Disease
Keywords: Inflammatory Bowel Disease; Coeliac Disease
MeSH Terms: conditions — Celiac Disease; Inflammatory Bowel Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Probiotic
- Probiotic (Experimental): Life Start Two
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Bifidobacterium infantis, 2 capsules (2.0E+9 CFU/capsule) 3 times/day for a total of 1.2E+10 CFU/day for 21 days.
  Other Names: Natren Inc.; Life Start Two; Bifidobacterium infantis

SUMMARY:
This exploratory study has been designed to determine the effect of the probiotic Bifidobacterium infantis vs. placebo orally administered over a period of 3 weeks on clinical features, Quality of Life parameters (QoL), intestinal permeability and inflammatory markers of patients having positive serological evidences of Celiac Disease.

DETAILED DESCRIPTION:
Objective: This exploratory study has been designed to determine the effect of the probiotic Bifidobacterium infantis vs. placebo orally administered over a period of 3 weeks on clinical features, Quality of Life parameters (QoL), intestinal permeability and inflammatory markers of patients having serological evidences of CD (positive serological markers). The testing period will be approximately three weeks between the results of serological testing and before the intestinal biopsy procedure during which time subjects are consuming a gluten-containing diet.

Study Design: A 3-weeks duration, placebo-controlled, double-blind, randomized study plan in ambulatory (non-hospitalized outpatients) patients, with 2 parallel groups. Treatment arms will be as follows:

A). Placebo 2 capsules 3 times daily (morning, evening and night).

B). Probiotics (Bifidobacterium infantis) 2 capsules 3 times per day (morning, evening and night).

ELIGIBILITY:
Inclusion Criteria:

* Signing the Informed consent.
* Men or women, 18-75 years old.
* BMI between 18.5 and 35.
* Patients shall have a positive CD-related serology (combined positivity of DGP/tTG Screen plus IgA anti-tTG and or IgA a-DGP tests).
* Patients will abstain from taking medications prohibited by the study from the 7 days prior the enrolment to the end of the trial: NSAIDs, aspirin, lactulose, probiotics and prebiotics in any form of administration (eg. Yogurts or other dairy products)..
* Alcohol consumption is prohibited during the same period.
* Patients should commit to attend on scheduled days, in accordance with the study calendar.
* To be interested in participating the trial

Exclusion Criteria:

* Patients with refractory CD or severe complications thereof, enteropathy-associated T-cell Lymphoma (EATL), ulcerative jejunitis, perforation, severe osteoporosis, malnutrition, among others.
* Individuals with symptoms suggestive of lymphoma or any other serious CD complication taking special care in recently-diagnosed patients, 50 years old or older, in whom EATL must be ruled out by standard methods.
* Individuals with other active chronic GI pathologies like Crohn's disease, ulcerative colitis and irritable bowel syndrome, microscopic colitis, and lactose intolerance.
* Patients with Type 1 or Type 2 diabetes or other autoimmune diseases, such as autoimmune hepatitis and primary biliary cirrhosis.
* Individuals with co-morbidities whose participation, in the investigator's judgment, would be inadvisable; for instance, unstable clinical conditions such as chronic obstructive pulmonary disease, angina pectoris, severe cardio-respiratory conditions, etc.
* Individuals with symptomatic neurological or psychiatric conditions that could potentially interfere with the study.
* Individuals with a clinical severity requiring immediate treatment at the consideration of the investigator.
* Patients with hemoglobin levels less than 8.5 g/dL or who had donated blood in the last 56 days or donated a unit of plasma in the last 7 days.
* Patients with a history of alcohol or drug abuse in the prior 2 years.
* Individuals taking "prohibited" medications in relation to the study (see point 6, previous section).
* Individuals with a history of neoplasia.
* Individuals participating in another clinical study that either involves medications or concluded during the last 30 days.
* Individuals previously exposed to Bifidobacteria species.
* Subjects not willing to maintain a gluten-containing diet during the 3-weeks period of the trial
* Pregnant women.
* Allergies to goat milk; no recent or planned dietary changes, esp. regarding gluten intake.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability changes | 21 days
  Subjects will come to the laboratory after an overnight fast, ingest the sugar probes, and collect all urine passed over the ensuing 24 hours into a pre-weighed container with 5 ml of 10% thymol in isopropanol. Urine will be vigorously mixed, total volume recorded, and aliquots rapidly frozen for subsequent transport and analysis. To evaluate intestinal permeability, subjects will ingest a solution containing: 5 g lactulose (Technilab, Montreal, Quebec, Canada), and 2 g mannitol (Sigma, St Louis, Missouri, USA) in 450 ml of water (osmolality approximately 1800 mOsmol/l).

SECONDARY OUTCOMES:
Changes in the cytokine profile. | 21 days
  Mononuclear cells obtained from blood will be isolated by Ficoll-Hypaque density centrifugation and resuspended in complete media/Dulbecco's modified Eagle medium. These mononuclear cells will be termed peripheral blood mononuclear cells (PBMCs). PBMCs will be incubated, nonstimulated, for 72 hours at 37°C in a 5% CO2 humidified atmosphere. Nonstimulated PBMC cytokine reflects the cytokine milieu from wich the PBMCs were originally isolated. Interleukin(IL)-10 and IL-12p40 cytokine levels will be measured using enzyme-linked immunosorbent assays.

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Bai, M.D., Study Director — Dr. C. Bonorino Udaondo Gastroenterology Hospital; Edgardo Smecuol, M.D., Principal Investigator — Dr. C. Bonorino Udaondo Gastroenterology Hospital
Locations (1):
- Dr. C. Bonorino Udanondo Gastroenterology Hospital, Buenos Aires, Argentina

REFERENCES:
- [Background] Sander GR, Cummins AG, Henshall T, Powell BC. Rapid disruption of intestinal barrier function by gliadin involves altered expression of apical junctional proteins. FEBS Lett. 2005 Aug 29;579(21):4851-5. doi: 10.1016/j.febslet.2005.07.066. PMID 16099460
- [Background] Maiuri L, Ciacci C, Ricciardelli I, Vacca L, Raia V, Rispo A, Griffin M, Issekutz T, Quaratino S, Londei M. Unexpected role of surface transglutaminase type II in celiac disease. Gastroenterology. 2005 Nov;129(5):1400-13. doi: 10.1053/j.gastro.2005.07.054. PMID 16285941
- [Background] Barone MV, Gimigliano A, Castoria G, Paolella G, Maurano F, Paparo F, Maglio M, Mineo A, Miele E, Nanayakkara M, Troncone R, Auricchio S. Growth factor-like activity of gliadin, an alimentary protein: implications for coeliac disease. Gut. 2007 Apr;56(4):480-8. doi: 10.1136/gut.2005.086637. Epub 2006 Aug 4. PMID 16891357
- [Background] Rollan G, De Angelis M, Gobbetti M, de Valdez GF. Proteolytic activity and reduction of gliadin-like fractions by sourdough lactobacilli. J Appl Microbiol. 2005;99(6):1495-502. doi: 10.1111/j.1365-2672.2005.02730.x. PMID 16313422
- [Background] Di Cagno R, De Angelis M, Lavermicocca P, De Vincenzi M, Giovannini C, Faccia M, Gobbetti M. Proteolysis by sourdough lactic acid bacteria: effects on wheat flour protein fractions and gliadin peptides involved in human cereal intolerance. Appl Environ Microbiol. 2002 Feb;68(2):623-33. doi: 10.1128/AEM.68.2.623-633.2002. PMID 11823200
- [Background] Di Cagno R, De Angelis M, Auricchio S, Greco L, Clarke C, De Vincenzi M, Giovannini C, D'Archivio M, Landolfo F, Parrilli G, Minervini F, Arendt E, Gobbetti M. Sourdough bread made from wheat and nontoxic flours and started with selected lactobacilli is tolerated in celiac sprue patients. Appl Environ Microbiol. 2004 Feb;70(2):1088-96. doi: 10.1128/AEM.70.2.1088-1096.2004. PMID 14766592
- [Background] Gerez CL, Rollan GC, de Valdez GF. Gluten breakdown by lactobacilli and pediococci strains isolated from sourdough. Lett Appl Microbiol. 2006 May;42(5):459-64. doi: 10.1111/j.1472-765X.2006.01889.x. PMID 16620203
- [Background] Rizzello CG, De Angelis M, Di Cagno R, Camarca A, Silano M, Losito I, De Vincenzi M, De Bari MD, Palmisano F, Maurano F, Gianfrani C, Gobbetti M. Highly efficient gluten degradation by lactobacilli and fungal proteases during food processing: new perspectives for celiac disease. Appl Environ Microbiol. 2007 Jul;73(14):4499-507. doi: 10.1128/AEM.00260-07. Epub 2007 May 18. PMID 17513580
- [Background] Lindfors K, Blomqvist T, Juuti-Uusitalo K, Stenman S, Venalainen J, Maki M, Kaukinen K. Live probiotic Bifidobacterium lactis bacteria inhibit the toxic effects induced by wheat gliadin in epithelial cell culture. Clin Exp Immunol. 2008 Jun;152(3):552-8. doi: 10.1111/j.1365-2249.2008.03635.x. Epub 2008 Apr 16. PMID 18422736
- [Background] De Palma G, Nadal I, Medina M, Donat E, Ribes-Koninckx C, Calabuig M, Sanz Y. Intestinal dysbiosis and reduced immunoglobulin-coated bacteria associated with coeliac disease in children. BMC Microbiol. 2010 Feb 24;10:63. doi: 10.1186/1471-2180-10-63. PMID 20181275
- [Background] De Palma G, Cinova J, Stepankova R, Tuckova L, Sanz Y. Pivotal Advance: Bifidobacteria and Gram-negative bacteria differentially influence immune responses in the proinflammatory milieu of celiac disease. J Leukoc Biol. 2010 May;87(5):765-78. doi: 10.1189/jlb.0709471. Epub 2009 Dec 10. PMID 20007908
- [Background] Di Cagno R, Rizzello CG, Gagliardi F, Ricciuti P, Ndagijimana M, Francavilla R, Guerzoni ME, Crecchio C, Gobbetti M, De Angelis M. Different fecal microbiotas and volatile organic compounds in treated and untreated children with celiac disease. Appl Environ Microbiol. 2009 Jun;75(12):3963-71. doi: 10.1128/AEM.02793-08. Epub 2009 Apr 17. PMID 19376912
- [Background] Collado MC, Donat E, Ribes-Koninckx C, Calabuig M, Sanz Y. Imbalances in faecal and duodenal Bifidobacterium species composition in active and non-active coeliac disease. BMC Microbiol. 2008 Dec 22;8:232. doi: 10.1186/1471-2180-8-232. PMID 19102766
- [Background] Medina M, De Palma G, Ribes-Koninckx C, Calabuig M, Sanz Y. Bifidobacterium strains suppress in vitro the pro-inflammatory milieu triggered by the large intestinal microbiota of coeliac patients. J Inflamm (Lond). 2008 Nov 3;5:19. doi: 10.1186/1476-9255-5-19. PMID 18980693
- [Background] Nadal I, Donant E, Ribes-Koninckx C, Calabuig M, Sanz Y. Imbalance in the composition of the duodenal microbiota of children with coeliac disease. J Med Microbiol. 2007 Dec;56(Pt 12):1669-1674. doi: 10.1099/jmm.0.47410-0. PMID 18033837
- [Derived] Smecuol E, Hwang HJ, Sugai E, Corso L, Chernavsky AC, Bellavite FP, Gonzalez A, Vodanovich F, Moreno ML, Vazquez H, Lozano G, Niveloni S, Mazure R, Meddings J, Maurino E, Bai JC. Exploratory, randomized, double-blind, placebo-controlled study on the effects of Bifidobacterium infantis natren life start strain super strain in active celiac disease. J Clin Gastroenterol. 2013 Feb;47(2):139-47. doi: 10.1097/MCG.0b013e31827759ac. PMID 23314670